CLINICAL TRIAL: NCT05005507
Title: A Phase 2, Open-label, Multicenter Study to Assess Efficacy, Safety, Tolerability, and Pharmacokinetics of Treatment With JNJ-73763989, Nucleos(t)Ide Analogs, and Pegylated Interferon Alpha-2a in Patients With Chronic Hepatitis B Virus Infection
Brief Title: A Study of JNJ-73763989, Pegylated Interferon Alpha-2a and Nucleos(t)Ide Analogs in Participants With Chronic Hepatitis B Virus Infection
Acronym: PENGUIN-2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A strategic decision was made to not further execute the study. This decision was not based on a safety concern.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109070; 2021-002450-81 (EudraCT Number); 73763989PAHPB2007 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-08-12; First posted 2021-08-13 (Actual); Results first posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-01

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: JNJ-73763989 + nucleos(t)ide analog (NA) + pegylated interferon alpha-2a (PegIFN-alpha-2a) (Experimental): Participants will receive JNJ-73763989 subcutaneous (SC) injection once every 4 weeks for 24 weeks plus NA treatment (either entecavir [ETV], tenofovir disoproxil or tenofovir alafenamide [TAF] tablets orally) once daily for 24 weeks plus PegIFN-alpha-2a SC injection once weekly for 24 weeks.
  Interventions: Drug: JNJ-73763989; Drug: PegIFN-alpha-2a; Drug: Tenofovir disoproxil; Drug: TAF; Drug: ETV
- Arm 2: JNJ-73763989 + NA + PegIFN-alpha-2a (Experimental): Participants will receive JNJ-73763989 SC injection once every 4 weeks for 24 weeks plus NA treatment (either ETV, tenofovir disoproxil, or TAF tablets orally) once daily for 24 weeks plus PegIFN-alpha-2a SC injection once weekly from Week 12 till Week 24.
  Interventions: Drug: JNJ-73763989; Drug: PegIFN-alpha-2a; Drug: Tenofovir disoproxil; Drug: TAF; Drug: ETV
- Arm 3: JNJ-73763989 + NA + PegIFN-alpha-2a (Experimental): Participants will receive JNJ-73763989 SC injection once every 4 weeks for 24 weeks plus NA treatment (either ETV, tenofovir disoproxil or TAF tablets orally) once daily for 24 weeks plus PegIFN-alpha-2a SC injection once weekly from baseline till Week 12.
  Interventions: Drug: JNJ-73763989; Drug: PegIFN-alpha-2a; Drug: Tenofovir disoproxil; Drug: TAF; Drug: ETV

INTERVENTIONS:
Drug: JNJ-73763989 — JNJ-73763989 will be administered subcutaneously once every 4 weeks.
  Other Names: JNJ-3989
Drug: PegIFN-alpha-2a — PegIFN-alpha-2a will be administered subcutaneously once weekly.
Drug: Tenofovir disoproxil — Tenofovir disoproxil film-coated tablet will be administered orally once daily.
Drug: TAF — TAF film-coated tablet will be administered orally once daily.
Drug: ETV — ETV film-coated tablet will be administered orally once daily.

SUMMARY:
The purpose of this study is to evaluate the efficacy in terms of hepatitis B surface antigen (HBsAg) changes from baseline for the treatment regimens of 24 weeks of JNJ-73763989 + 24 weeks of nucleos(t)ide analog (NA) + 12 or 24 weeks of pegylated interferon alpha-2a (PegIFN-alpha-2a) (with immediate or delayed start of PegIFN-alpha-2a treatment).

DETAILED DESCRIPTION:
JNJ-73763989 (JNJ-3989) is a liver-targeted antiviral therapeutic for subcutaneous injection designed to treat chronic hepatitis B virus (HBV) infection via a ribonucleic acid interference (RNAi) mechanism. Combination treatment with JNJ-73763989 and NA has the potential to specifically decrease HBV viral antigen levels and inhibit viral replication. Since HBsAg is immune suppressive, the direct reduction of HBsAg levels by JNJ-73763989 is anticipated to contribute to the restoration of the immune response that is impaired in chronic HBV infection. Pegylated interferon (PegIFN) is an approved drug for the treatment of chronic HBV infection and after a finite treatment duration of 48 weeks results in slightly increased HBsAg seroclearance rates. The primary hypothesis of this study is that at least one of the combination regimens of JNJ-73763989+NA+PegIFN-alpha-2a is more efficacious than NA treatment alone (standard of care), as measured by the primary efficacy endpoint. This study will be conducted in 3 periods: Screening Period (4 weeks), Treatment Period (24 weeks) and Follow-up (FU) Period (48 weeks), starting at Week 24. Safety assessments will include adverse events (AEs), serious AEs, clinical safety laboratory tests, electrocardiograms (ECGs), vital signs, ophthalmologic examinations and physical examinations. Total duration of individual participation will be up to 76 weeks (including screening period).

ELIGIBILITY:
Inclusion Criteria:

* Medically stable based on physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening
* Participants must have a body mass index between 18.0 and 35.0 kilograms per meter square (kg/m^2) inclusive
* Participants with chronic hepatitis B who should: a) be chronic hepatitis B e antigen (HBeAg) -negative; b) be anti-HBe antibody-positive; c) be currently receiving nucleos(t)ide analog (NA) treatment for at least 2 years prior to screening; d) have serum hepatitis B virus (HBV) deoxyribonucleic acid (DNA) less than (<) 60 international unit/milliliter (IU/mL) on 2 sequential measurements at least 6 months apart; e) have alanine aminotransferase (ALT) values < 2.0x upper limit of normal (ULN) on 2 sequential measurements at least 6 months apart
* Hepatitis B surface antigen (HBsAg) greater than (>) 5 IU/mL at screening
* Fibroscan liver stiffness measurement less than or equal to (<=) 9.0 kilopascal (kPa) within 6 months prior to screening

Exclusion Criteria:

* History or signs of cirrhosis or portal hypertension
* Evidence of hepatitis A, C, D, E virus infection, or human immunodeficiency virus (HIV) infection
* Liver disease of non-HBV etiology
* Clinically relevant alcohol or drug abuse within 12 months of screening
* Participants who meet any of the additional exclusion criteria for pegylated interferon alpha-2a (PegIFN- α2a) as described in local prescribing information (example, refer to Pegasys SmPC or Pegasys USPI) per the investigator's discretion. Key exclusion criteria for PegIFN- α2a include: a) Participants with signs or symptoms compatible with autoimmune disorders. b) Participants with bone marrow suppression. c) Participants with hypoglycaemia, hyperglycaemia, and/or diabetes mellitus, who cannot be effectively controlled by medication. d) Participants with pre-existing ophthalmologic disorders. e) Participants with one or more of the following laboratory abnormalities: i) Absolute neutrophil count less than (<)1,500 cells/mm3 (<1,000 cells/mm³ for black or African American participants). ii) Serum creatinine >1.5x ULN. iii) Inadequately controlled thyroid function (thyroid stimulating hormone [TSH] and thyroxine [T4]). f) Participants with a history of a severe psychiatric disorder including severe depression, suicidal ideation and attempted suicide, or a current depression or other psychiatric disorder that is not adequately controlled on a stable medication regimen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (12):
- I.D. Care, Inc., Hillsborough, New Jersey, United States
- Canada (2):
  - Vancouver ID Research and Care Centre Society, Vancouver, British Columbia
  - GI Research Institute (G.I.R.I.), Vancouver, British Columbia
- Kagawa Prefectural Central Hospital, Takamatsu, Japan
- Poland (3):
  - PUNKT ZDROWIA Hlebowicz Jakubowski Lekarze sp.p., Gdansk
  - ID Clinic, Mysłowice
  - EMC Instytut Medyczny SA, Wroclaw
- Spain (4):
  - Hosp. Univ. Vall D Hebron, Barcelona
  - Hosp. Univ. Infanta Leonor, Madrid
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Alvaro Cunqueiro, Vigo
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical- trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only 1 participant was enrolled in the study in Arm 1: JNJ-73763989 + nucleos(t)ide analog (NA) + pegylated interferon alpha-2a (PegIFN-alpha-2a) but did not complete the study. Participants were also planned to be enrolled in Arms 2 and 3 but were not enrolled as the study terminated prematurely based on a strategic decision and not for safety reasons.
Groups:
- Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a: Participants received JNJ-73763989 200 milligrams (mg) subcutaneous (SC) injection on Day 1 plus NA treatment (entecavir [ETV] 0.5 mg tablet) orally once daily from Day 1 to Day 16 plus pegylated interferon alpha-2a (PegIFN-alpha-2a) 180 micrograms (mcg) SC injection on Days 1, 8, and 15.
Period: Overall Study
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Started | 1
Completed | 0
Not Completed | 1
Not completed — Premature termination of study | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (NA) — Standard deviation could not be calculated for 1 participant.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Reduction of at Least 2log10 International Units Per Milliliter (IU/mL) in Hepatitis B Surface Antigen (HBsAg) Levels From Baseline at Week 24 (End of Study Intervention [EOSI])
Description: Percentage of participants with a reduction of at least 2log10 IU/mL in HBsAg levels from baseline at Week 24 (EOSI) were planned to be reported.
Time Frame: Week 24
Population: Full analysis set (FAS) included all participants who were randomly assigned to an intervention arm in the intervention-specific appendix (ISA) and received at least 1 dose of study intervention. The data was not collected and analyzed for this outcome measure due to premature termination of the study.
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 0

2. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Up to 1 month 26 days
Population: Safety analysis set included all participants who received at least 1 dose of study intervention within the ISA.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 1
Percentage of participants | 0

3. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE is any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: Up to 1 month 26 days
Population: Safety analysis set included all participants who received at least 1 dose of study intervention within the ISA.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 1
Percentage of participants | 0

4. Secondary Outcome: Percentage of Participants With Abnormalities in Clinical Laboratory Tests
Description: Percentage of participants with abnormalities in clinical laboratory tests including hematology, blood coagulation, blood biochemistry, urinalysis, urine chemistry, renal biomarkers, were reported.
Time Frame: Up to 1 month 26 days
Population: Safety analysis set included all participants who received at least 1 dose of study intervention within the ISA.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 1
Percentage of participants
  Hematology | 0
  Blood coagulation | 0
  Blood biochemistry | 0
  Urinalysis | 0
  Urine chemistry | 0
  Renal biomarker | 0

5. Secondary Outcome: Percentage of Participants With Abnormalities in 12-Lead Electrocardiograms (ECGs)
Description: Percentage of participants with abnormalities in 12-Lead ECGs were reported.
Time Frame: Up to 1 month 26 days
Population: Safety analysis set included all participants who received at least 1 dose of study intervention within the ISA.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 1
Percentage of participants | 0

6. Secondary Outcome: Percentage of Participants With Abnormalities in Vital Signs
Description: Percentage of participants with abnormalities in vital signs were reported.
Time Frame: Up to 1 month 26 days
Population: Safety analysis set included all participants who received at least 1 dose of study intervention within the ISA.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 1
Percentage of participants | 0

7. Secondary Outcome: Percentage of Participants With Abnormalities in Ophthalmologic Examination
Description: Percentage of participants with abnormalities in ophthalmologic examination were planned to be reported.
Time Frame: Weeks 8 and 20
Population: Safety analysis set included all participants who received at least 1 dose of study intervention within the ISA. The data was not collected and analyzed for this outcome measure due to premature termination of the study.
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 0

8. Secondary Outcome: Percentage of Participants With Abnormalities in Physical Examination
Description: Percentage of participants with abnormalities in physical examination were planned to be reported.
Time Frame: Week 24
Population: as for outcome 7
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 0

9. Secondary Outcome: Percentage of Participants Meeting the Protocol-defined Nucleos(t)Ide Analog (NA) Treatment Completion Criteria Based on the Week 24 (EOSI) or Follow-up Week 2 Visits
Description: Percentage of participants meeting the protocol-defined NA treatment completion criteria based on the Week 24 (EOSI) or follow-up Week 2 visits was planned to be reported. NA treatment completion criteria were as follows: (a) participant had alanine transaminase (ALT) <3*upper limits of normal (ULN); (b) participant had Hepatitis B Virus (HBV) Deoxyribonucleic acid (DNA) <20 international units per milliliter (IU/mL); (c) participant was Hepatitis B e antigen (HBeAg)-negative; (d) participant had Hepatitis B surface antigen (HBsAg<10 IU/mL.
Time Frame: Week 24 (EOSI) and follow-up Week 2
Population: FAS included all participants who were randomly assigned to an intervention arm in the ISA and received at least 1 dose of study intervention. The data was not collected and analyzed for this outcome measure due to premature termination of the study.
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 0

10. Secondary Outcome: Percentage of Participants With HBsAg Seroclearance at Follow-up Weeks 24 and 48 Without Re-starting NA Treatment
Description: Percentage of participants with HBsAg seroclearance at follow-up Weeks 24 and 48 without re-starting NA treatment were planned to be reported. Seroclearance of HBsAg is defined as a (quantitative) HBsAg level <lower limit of quantitation (LLOQ). LLOQ is 0.05 International Units per milliliter (IU/mL).
Time Frame: Follow-up Weeks 24 and 48
Population: as for outcome 9
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 0

11. Secondary Outcome: Percentage of Participants With Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) < (Less Than) LLOQ at Follow-up Weeks 24 and 48 Without Re-starting NA Treatment
Description: Percentage of participants with HBV DNA <LLOQ at follow-up Weeks 24 and 48 without re-starting NA treatment were planned to be reported. LLOQ is 0.05 IU/mL.
Time Frame: Follow-up Weeks 24 and 48
Population: as for outcome 9
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 0

12. Secondary Outcome: Percentage of Participants With Virologic Flares
Description: Percentage of participants with virologic flares were reported. The start of a confirmed virologic flare is defined as the first date of two consecutive visits with HBV DNA >200 IU/mL. The end date of the same confirmed virologic flare is defined as the first date when HBV DNA value returns to less than or equal to (<=)200 IU/mL or the date of NA treatment restart, whichever comes first.
Time Frame: Up to 1 month 26 days
Population: FAS included all participants who were randomly assigned to an intervention arm in the ISA and received at least 1 dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 1
Percentage of participants | 0

13. Secondary Outcome: Percentage of Participants With Biochemical Flares
Description: Percentage of participants with biochemical flares were reported. The start date of a confirmed off-treatment biochemical flare: the first date of two consecutive visits with ALT and/or AST>=3x ULN and >=3x off-treatment/on-treatment nadir (that is, lowest value observed during off-treatment period up to the time point of meeting the biochemical flare criteria) while the participant does not receive any of the study interventions. The end date of the same off-treatment/on-treatment biochemical flare: the first date when there is a 50% reduction from the peak ALT and/or AST level & <3x ULN.
Time Frame: Up to 1 month 26 days
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 1
Percentage of participants | 0

14. Secondary Outcome: Percentage of Participants Requiring Nucleos(t)Ide Analog (NA) Re-treatment
Description: Percentage of participants requiring NA re-treatment were planned to be reported.
Time Frame: Up to 72 weeks
Population: as for outcome 9
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 0

15. Secondary Outcome: Percentage of Participants With HBsAg, Hepatitis B e Antigen (HBeAg), HBV DNA, and Alanine Aminotransferase (ALT) Levels Below/Above Different Cut-offs
Description: Percentage of participants with HBsAg, HBeAg, HBV DNA, and ALT levels below/above different cut-offs were planned to be reported.
Time Frame: Up to 72 weeks
Population: as for outcome 9
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 0

16. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion
Description: Percentage of participants with HBsAg seroconversion were planned to be reported. Seroconversion of HBsAg is defined as having achieved HBsAg seroclearance (quantitative HBsAg level <LLOQ) and appearance of anti-HBs antibodies. LLOQ is 0.05 IU/mL.
Time Frame: Up to 72 weeks
Population: as for outcome 9
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 0

17. Secondary Outcome: Change From Baseline in HBsAg Over Time
Description: Change from baseline in HBsAg over time were planned to be reported.
Time Frame: Baseline up to Week 72
Population: as for outcome 9
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 0

18. Secondary Outcome: Time to Achieve HBsAg Seroclearance
Description: Time to achieve HBsAg seroclearance were planned to be reported. Time to achieve HBsAg seroclearance is defined as the number of days between the date of first study intervention intake and the date of the first occurrence of HBsAg seroclearance (that is, the date of the first HBsAg seroclearance - the date of first study intervention intake + 1). Seroclearance of HBsAg is defined as a (quantitative) HBsAg level <LLOQ. LLOQ is 0.05 IU/mL.
Time Frame: Up to 72 weeks
Population: as for outcome 9
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 0

19. Secondary Outcome: Time to Achieve HBsAg Seroconversion
Description: Time to achieve HBsAg seroconversion were planned to be reported. Time to achieve HBsAg seroconversion is defined as the number of days between the date of first study intervention intake and the date of the first occurrence of HBsAg seroclearance and appearance of anti-HBs antibodies (that is, the date of the first HBsAg seroclearance and anti-HBs antibodies - the date of first study intervention intake + 1). Seroconversion of HBsAg is defined as having achieved HBsAg seroclearance (quantitative HBsAg level <LLOQ) and appearance of anti-HBs antibodies. LLOQ is 0.05 IU/mL.
Time Frame: Up to 72 weeks
Population: as for outcome 9
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 0

20. Secondary Outcome: Time to Achieve HBV DNA <Lower Limit of Quantitation (LLOQ)
Description: Time to achieve HBV DNA <LLOQ were planned to be reported. Time to achieve HBV DNA <LLOQ is defined as the number of days between HBV DNA >LLOQ for participants who re-treated with NA and the date of the first occurrence of HBV DNA < LLOQ after NA re-treatment (that is, the date of the HBV DNA < LLOQ after being re-treated with NA - the date of first occurrence of HBV DNA>LLOQ + 1). LLOQ is 0.05 IU/mL.
Time Frame: Up to 72 weeks
Population: as for outcome 9
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 0

21. Secondary Outcome: Percentage of Participants With Virologic Breakthrough
Description: Percentage of participants with virologic breakthrough were planned to be reported. HBV virological breakthrough is defined as having a confirmed on-treatment HBV DNA increase by >1 log10 from nadir level (lowest level reached during treatment) in participants who did not have on-treatment HBV DNA level below the LLOQ or a confirmed on-treatment HBV DNA level >200 IU/mL in participants who had on-treatment HBV DNA level below the LLOQ. LLOQ is 0.05 IU/mL.
Time Frame: Up to Week 24
Population: as for outcome 9
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 0

22. Secondary Outcome: Serum Concentration of JNJ-73763989 (JNJ-73763924 and JNJ-73763976)
Description: Serum concentration of JNJ-73763989 (JNJ-73763924 and JNJ-73763976) were planned to be reported.
Time Frame: Up to 72 weeks
Population: Pharmacokinetics (PK) analysis set included all participants who received at least 1 dose of study intervention and have at least 1 valid blood sample drawn for PK analysis. The data was not collected and analyzed for this outcome measure due to premature termination of the study.
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 0

23. Secondary Outcome: Serum Concentration of Nucleos(t)Ide Analog (NA) (Entecavir [ETV])
Description: Serum concentration of NA (ETV) was planned to be reported.
Time Frame: Up to 72 weeks
Population: PK analysis set included all participants who received at least 1 dose of study intervention and have at least 1 valid blood sample drawn for PK analysis. The data was not collected and analyzed for this outcome measure due to premature termination of the study.
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 0

24. Secondary Outcome: Serum Concentration of PegIFN-alpha-2a
Description: Serum concentration of PegIFN-alpha-2a was planned to be reported.
Time Frame: Up to 72 weeks
Population: as for outcome 23
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 1 month 26 days
Description: Safety analysis set included all participants who received at least 1 dose of study intervention within this intervention-specific appendix (ISA). Participants were analyzed according to the study intervention they actually received.
Arm/Group | Arm 1: JNJ-73763989+Nucleos(t)Ide Analog (NA)+PegIFN-alpha-2a
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Only 1 participant was enrolled in the study in Arm 1. Participants were also planned to be enrolled in Arms 2 and 3 but were not enrolled as the study terminated prematurely based on a strategic decision and not for safety reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT05005507/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT05005507/SAP_001.pdf